CLINICAL TRIAL: NCT02938689
Title: Efficacy Comparison of the Exercises Based on the Lumbar Extension and Flexion in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sun Gun Chung, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNUH-1607-199-782
Record Dates: First submitted 2016-10-11; First posted 2016-10-19 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Lumbar extension exercise (Experimental): Exercise education based on Mckenzie lumbar extension exercise for 4 weeks
  Interventions: Other: Exercise
- Lumbar flextion exercise (Active Comparator): Exercise education based on Wilillams lumbar flexion exercise for 4 weeks
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise

SUMMARY:
This study is to compare the efficacy of exercises based on the lumbar extension and flexion on the pain relief and the prevention of pain recurrence in chronic low back pain patients.

DETAILED DESCRIPTION:
68 people that meet the inclusion criteria on screening test are assigned to one of two groups by randomization. Each of the group learns one of the exercises based on the lumbar extension or flexion for four weeks. The main outcome variables are measured and compared respectively in baseline, immediately after the education, 3, 6, 12 months after the enrollment. Finally lumbar extension exercise is verified whether it is more effective than the lumbar flexion exercise on the pain relief and the prevention of pain recurrence in chronic low back pain patients.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain (>6 months, VAS score of 5 or above)
* presence of discogenic or axial pain
* duration of >6 months

Exclusion Criteria:

* Spondylolisthesis or retrolisthesis on radiograph
* Hx of spine surgery
* Hx of any spine intervention within 3 months
* other neurological, inflammatory, or poor medical conditions
* who cannot understand or conduct the protocol of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Average Back pain VAS score (0~10) at 12 month | Baseline, Month 1, Month 3, Month 6, Month 12
  Describe the degree of pain by VAS score

SECONDARY OUTCOMES:
brief pain inventory (right now pain, worst pain, least pain, pain interference) | Baseline, Month 1, Month 3, Month 6, Month 12
  Describe the degree of pain by survey
Oswestry Disability Questionnaire | Baseline, Month 1, Month 3, Month 6, Month 12
  Describe the degree of pain by survey
EQ-5D | Baseline, Month 1, Month 3, Month 6, Month 12
  Describe the health-related quality of life
PASE | Baseline, Month 1, Month 3, Month 6, Month 12
  Describe the status of physical activity
How often did the subject conduct exercise in the past a month? (5 levels) | Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 12
  1. 3 times or more a day
  2. once or twice a day
  3. 4 times or more a week, but less than once a day
  4. 1-3 times a week
  5. less than once a week

CONTACTS AND LOCATIONS:
Overall Officials: Sun Gun Chung, MD. PhD, Study Chair — Department of Rehabilitation Medicine, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park CH, Beom J, Chung CK, Kim CH, Lee MY, Park MW, Kim K, Chung SG. Long-term effects of lumbar flexion versus extension exercises for chronic axial low back pain: a randomized controlled trial. Sci Rep. 2024 Feb 1;14(1):2714. doi: 10.1038/s41598-024-51769-2. PMID 38302483